CLINICAL TRIAL: NCT05434910
Title: Study Protocol: The Effect of Blood Pressure on Cerebral Blood Flow in Comatose Out-of-hospital Cardiac Arrest Patients
Brief Title: Blood Pressure and Cerebral Blood Flow After Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Niels Damkjær Olesen (Other)
Responsible Party: Sponsor-Investigator, Niels Damkjær Olesen, Principal investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-22000181
Record Dates: First submitted 2022-06-16; First posted 2022-06-28 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Post-Cardiac Arrest Syndrome
Keywords: Out-Of-Hospital Cardiac Arrest; Blood pressure; Cerebral blood flow; Cerebral metabolism; Cardiac output; Noradrenaline; Post-Cardiac Arrest Syndrome
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Post-Cardiac Arrest Syndrome | interventions — Arterial Pressure

STUDY DESIGN:
Intervention Model Description: In the study, the infusion rate of noradrenaline will be temporarily adjusted to the following three levels MAP: 65, 80, and 95 mmHg and measurements will be conducted at each level of MAP. See detailed description elsewhere.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Changes in mean arterial pressure (MAP).
  In all subjects MAP is temporally adjusted using noradrenaline to the following three levels:
  * MAP 65 mmHg.
  * MAP 80 mmHg.
  * MAP 95 mmHg. When MAP has been stable at the given level for 20 min, measurements are conducted over 5 min. When the measurements are done, the study is finished. The study will last approximately 2 hours.
  Measurements include internal carotid and vertebral artery blood flow, mean arterial pressure, heart rate, peripheral O2 saturation, cardiac output, left ventricle ejection fraction, frontal lobe and muscle oxygenation, blood velocity in the middle cerebral artery, pupillometry, and arterial, central venous, and internal jugular venous gas variables and blood samples for analysis of metabolomics.
  Interventions: Other: Changes in mean arterial pressure

INTERVENTIONS:
Other: Changes in mean arterial pressure — MAP set at 65 mmHg for 25 min by infusion of noradrenaline. MAP set at 80 mmHg for 25 min by infusion of noradrenaline. MAP set at 95 mmHg for 25 min by infusion of noradrenaline.

SUMMARY:
Comatose patients that are admitted to an intensive care unit after out-of-hospital cardiac arrest (OCHA) have a high mortality, particularly due to hypoxic-ischemic neurologic injury. These patients often require vasopressors to maintain mean arterial pressure (MAP), but it is unclear what level of MAP should be aimed for. The objective of the study is to evaluate whether cerebral blood flow (CBF) and cerebral metabolism can be increased by maintaining MAP at a higher level than that used in clinical practice. The study will include twenty comatose patients within two days following resuscitation after OCHA. In the study, MAP is adjusted by infusion of noradrenaline, to a low, moderate, and high level for a short time. The low level of MAP used in the study, corresponds to the level aimed for in clinical practice. The CBF will be evaluated on the neck using ultrasound.

DETAILED DESCRIPTION:
Background Patients suffering out-of-hospital cardiac arrest (OCHA) have poor prognosis, and of the patients admitted to a hospital after return of spontaneous circulation, the 1 year survival is approximately 50% or lower. Anoxia during cardiac arrest and the subsequent reperfusion after resuscitation, affects the brain and other organs, and for patients admitted to an intensive care unit, the most frequent cause of death is hypoxic-ischemic brain injury. In the minutes after resuscitation, cerebral blood flow (CBF) increases markedly whereafter CBF is often reduced in the following 12 to 24 hours with regional differences whereby blood flow to some brain regions may be markedly reduced.

Mean arterial pressure (MAP) and cardiac output are often reduced following cardiac arrest due to myocardial dysfunction caused by ischemia-reperfusion injury, possible myocardial infarction that may have triggered the cardiac arrest, preexisting cardiac disease, and further, many patients develop a sepsis-like inflammatory response. Comatose survivors after cardiac arrest are generally cooled, intubated, and sedated using propofol that both lowers MAP and approximately halves both CBF and cerebral metabolic rate. Traditionally, CBF has been considered to be unaffected by changes in MAP between 60 to 150 mmHg by so-called cerebral autoregulation. Yet, CBF may be influenced by changes within this range of MAP and cerebral autoregulation is reported to be impaired in patients resuscitated after cardiac arrest whereby CBF becomes dependent on MAP.

Only limited data is available on the effect of MAP on CBF in OHCA patients. Cerebral oxygenation, as determined by near-infrared spectroscopy (NIRS), is unaffected by an increase in MAP from 65 to 85 mmHg using noradrenaline. However, evaluation of cerebral oxygenation using NIRS is affected by noradrenaline due to cutaneous vasoconstriction. In a similar study in anesthetized patients undergoing surgery, NIRS determined cerebral oxygenation was unaffected by an increase in MAP from 62 to 82 mmHg using noradrenaline whereas CBF increased by 15%.

Patients resuscitated after cardiac arrest are often hypotensive (generally defined as MAP < 60-65 mmHg) and hypotension is associated to poor neurologic outcome which may relate to reduced CBF and a larger degree of hypoxic-ischemic brain injury. It remains unclear, however, whether an increase in MAP using vasopressors such as noradrenaline, improves clinical outcome. Two small studies did not demonstrate any clear effect of maintaining MAP at 80-100 mmHg as compared to 65-75 mmHg on radiographic measurements or on biomarkers of neuronal damage. In clinical practice, a MAP of ≥ 65 mmHg is often aimed for, but it is unclear whether CBF and its metabolism may be increased by maintaining MAP at a higher level.

The study will include twenty comatose patients resuscitated after OCHA, due to a suspected or confirmed cardiac cause, and will be conducted within 2 days after resuscitation. The study will evaluate whether CBF and cerebral metabolism is affected by a short term increase in MAP to a level higher than that aimed for in clinical practice. MAP will be adjusted to 65, 80, and 95 mmHg in random order. Noradrenaline will be used as a tool to evaluate the effect of MAP as it has no direct effect on CBF.

Objective The purpose of the study is to evaluate whether CBF and cerebral metabolism is increased by maintaining MAP at a higher level than that used in clinical practice, in comatose patients following OHCA.

Hypotheses An increase in MAP from 65 to 95 mmHg will increase CBF and cerebral metabolism.

Methods

The study is a single-center, prospective cohort study of twenty consecutive patients that are comatose after resuscitation from OHCA. Patients will be included within 48 hours after resuscitation from OHCA but at the earliest 6 hours after return of spontaneous circulation. The experiment will be conducted at the earliest time possible after patient enrollment. The patients will be admitted to the Cardiologic Intensive Care Unit 2143 at Rigshospitalet, Copenhagen, Denmark. As part of routine care, patients are sedated using propofol, and noradrenaline is administered to maintain a MAP of 65 mmHg. It is estimated that more than 90% of the patients will require noradrenaline to maintain MAP. Before initiation of the study, the patient must have been hemodynamically stable for at least one hour, with a MAP of about 65 mmHg, and any changes in noradrenaline infusion may not exceed 25% of the dose during that time. Further, the sedation of the patient has to have been stable for at least 30 min and the end-tidal CO2 tension should be stable within 4.5 to 6.0 kPa. In the study, the investigators will temporarily adjust the infusion rate of noradrenaline to the following three levels MAP:

* MAP 65 mmHg.
* MAP 80 mmHg.
* MAP 95 mmHg.

The order of the three levels of MAP is randomized by drawing an envelope just before the start of the experiment. Administration of noradrenaline is by a central venous catheter, using an electronic infusion pump, and infusion speed is adjusted slowly until the given level of MAP is reached. Noradrenaline is short lasting and have no direct effect on CBF. When MAP has been stable at the given level for at least 20 min, measurements are conducted during the following 5 min, whereafter the infusion rate of noradrenaline is adjusted to the next level of MAP. If MAP does not drop to 65 mmHg by reducing or halting the infusion of noradrenaline, the evaluation is not conducted. No attempt will be made to reduce MAP (e.g. by administration of a vasodilator). If a noradrenaline infusion rate of > 0.5 µg/kg/min is needed to reach a given level of MAP, the infusion rate will not be increased further, and no evaluation will be conducted at that level or any higher levels of MAP. When measurements have been conducted at the three levels of MAP, or at the levels of MAP that were possible to evaluate, the study is complete, whereafter control of MAP will be according to clinical practice. The study will last for approximately two hours and will not influence patient care in any other respects. Patients that receive inotropes, including dopamine, dobutamine or milrinone apart from noradrenaline, as part of clinical practice, can be included in the study. The study is not an investigation of medicinal products as noradrenaline is used as a tool to control MAP.

Measurements

As part of clinical practice, an arterial line and a Swan-Ganz catheter are placed, lead II EKG and peripheral pulse oximetry are monitored and echocardiography is done. In the study, the following measurements are conducted:

* MAP is evaluated invasively by an arterial line.
* Heart rate by lead II EKG.
* Peripheral O2 saturation by pulse oximetry on a finger.
* Cardiac output and central venous pressure by Swan-Ganz catheter.
* Left ventricle ejection fraction by echocardiography.
* Guided by ultrasound, a catheter is placed in the internal jugular vein and the tip advanced retrogradely to the bulb of the vein in order to evaluate cerebral metabolism by comparing blood samples from the arterial line and the jugular venous blood that has passed the brain (see below).
* Blood is sampled from the arterial, Swan-Ganz, and jugular venous catheters for evaluation of hemoglobin, lactate, glucose, and bicarbonate concentration, pH, and O2 and CO2 tension by gas analysis.
* From the arterial and jugular venous catheters, blood will be sampled for analysis of metabolomics, i.e. a large number of metabolites in order to describe the metabolism of the body and the brain. In total, 63 ml of blood will be sampled.
* Blood flow in the internal carotid and vertebral arteries will be evaluated on the neck using duplex ultrasound with a linear probe. The internal carotid artery is insonated at least 1.5 cm distal to its bifurcation and the vertebral artery between the transverse processes C2-5 with the head turned approximately 30⁰ to the contralateral side. In order to limit the influence of ventilation, three recordings of approximately 15 s are conducted at each level of MAP and the mean is reported. A frequency of 8-12 MHz is used and gain is set as high as possible while vessel lumen is echo-free. Blood flow is calculated from the measured blood velocity and vessel diameter as evaluated using automatic software to track the vessel wall. The CBF is estimated as two times the sum of internal carotid and vertebral artery blood flow. Internal carotid and vertebral artery blood flow will also be corrected for any changes in PaCO2 using a factor of 19%/kPa (unpublished results from the study "Cerebral Blood Flow During Propofol Anaesthesia" NCT02951273).
* Cerebral and deltoid muscle oxygenation is evaluated using NIRS by placing an apparatus that emit and receive light on the forehead and the deltoid muscle, respectively.
* Blood velocity in the middle cerebral artery is evaluated by transcranial Doppler by placement of an ultrasound probe over the temple.
* Neuroptics NPi-200 pupillometry will be used to evaluate pupil size and light reaction.

Values are averaged over 2 min. Placement of a catheter in the internal jugular vein, evaluations using ultrasound and NIRS, pupillometry, and the blood samples are conducted as a part of the study. Study data will include hemodynamic measurements, physiological data, medicine administration, ventilator settings, and the results of blood samples taken as part of the study. Medical history will be assessed from the patient chart in regards to the inclusion and exclusion criteria and include age, gender, prior diseases, cause of cardiac arrest, prehospital and in-hospital treatment. Information on patient death or neurologic function upon hospital discharge will be recorded from the medical chart.

Statistics Trial size: The minimal clinically important difference in internal carotid artery blood flow between evaluations at MAP 65 and 95 mmHg is estimated to be 15%. A power calculation indicated that at least 16 patients were required to detect a difference in internal carotid artery blood flow of 15% corresponding to about 24 ml/min with a standard deviation for the change of 31 ml/min in order to obtain a 5% significance level and a power of 80%. The study will include 20 patients.

Ethics The study protocol (H-22000181) is approved by the Regional Ethical Committee of the Copenhagen Region (De Videnskabsetiske Komiteer Region Hovedstaden, 0045 38666395, Email: vek@regionh.dk, Address: Blegdamsvej 60. 1. sal opgang 94A11, DK-2100 Copenhagen, Denmark). Patients are comatose whereby they can not provide informed consent upon enrollment. Informed consent will be obtained from the next of kin and from another doctor at the hospital who is not affiliated with the department of cardiology or the treatment of the patient (legal guardian). The study will be stopped and the patient excluded, in case the next of kin or the legal guardian withdraws the consent to participate, if the patient is not in a condition to participate in the study, or if there is a suspicion of a complication related to the study. If the patient regains consciousness, he or she will be informed of the study and will have to provide informed consent in order to be included in the data set.

Patients will be deeply sedated and thus, will not experience any discomfort related to the study. The evaluations using ultrasound, NIRS, and pupillometry are without any risks. Placement of a catheter in the internal jugular vein is associated with a minor risk of bleeding and infection. The investigators consider that there is no increased risk by a short term increase in MAP to 80 and 95 mmHg. The study is monitored by the Danish Data Protection Agency.

The investigators have no conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are resuscitated within the last 48 hours after OCHA due to suspected or confirmed cardiac cause.
* Comatose or sedated (Glasgow Coma Score < 8 whereby the patient is unable to follow verbal commands).
* Age 18-90 years.

Exclusion Criteria:

* Patients that have had in-hospital cardiac arrest.
* Pregnancy, human chorionic gonadotropin is routinely measured in women < 60 years of age.
* Known hemorrhagic diathesis (medically induced coagulopathy due to blood thinners is not an exclusion criteria, except for those mentioned below).
* Anticoagulant therapy by warfarin with an INR > 2, Direct-Acting Oral Anticoagulants, or Eptifibatid.
* Suspected or confirmed stroke.
* Non-witnessed cardiac arrest with asystole as the initial rhythm.
* Known treatment limitation plan or a decision not to resuscitate the patient in case of a new cardiac arrest.
* Previous disease that makes 180 day survival unlikely.
* Known Cerebral Performance Category score 3 to 4 prior to cardiac arrest.
* Systolic blood pressure < 80 mmHg despite optimal fluid-, vasopressor-, and inotropic treatment.
* The need of noradrenaline infusion exceeding 0.3 μg/kg*min in order to maintain a MAP of 65 mmHg.
* Mechanical cardiac support devices.
* Known vascular disease in the internal carotid artery.
* Lack of visualization of the internal carotid artery, e.g. due to high placement of the bifurcation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in internal carotid artery blood flow. | Evaluations at 2 time points; when MAP is set to 65 and 95 mmHg. The evaluations are separated by approximately 30-60 min.
  Change in internal carotid artery blood flow [ml/min] as evaluated by duplex ultrasound when MAP is set to 65 and 95 mmHg.

SECONDARY OUTCOMES:
Change in cerebral blood flow. | Evaluations at 2 time points; when MAP is set to 65 and 95 mmHg. The evaluations are separated by approximately 30-60 min.
  Change in cerebral blood flow (two times internal carotid and vertebral artery blood flow) [ml/min] as evaluated by duplex ultrasound when MAP is set to 65 and 95 mmHg.
Change in vertebral artery blood flow. | Evaluations at 2 time points; when MAP is set to 65 and 95 mmHg. The evaluations are separated by approximately 30-60 min.
  Change in vertebral artery blood flow [ml/min] as evaluated by duplex ultrasound when MAP is set to 65 and 95 mmHg.
Change in arterial to internal jugular venous O2 content difference. | Blood is sampled 2 time points; when MAP is set to 65 and 95 mmHg. The evaluations are separated by approximately 30-60 min.
  Change in arterial to internal jugular venous O2 content difference [mM] as evaluated by blood gas analysis when MAP is set to 65 and 95 mmHg.
Change in arterial to internal jugular venous lactate concentration difference. | Blood is sampled 2 time points; when MAP is set to 65 and 95 mmHg. The evaluations are separated by approximately 30-60 min.
  Change in arterial to internal jugular venous lactate concentration difference [mM] as evaluated by blood gas analysis when MAP is set to 65 and 95 mmHg.
Change in arterial to internal jugular venous glucose concentration difference. | Blood is sampled 2 time points; when MAP is set to 65 and 95 mmHg. The evaluations are separated by approximately 30-60 min.
  Change in arterial to internal jugular venous glucose concentration difference [mM] as evaluated by blood gas analysis when MAP is set to 65 and 95 mmHg.
Change in cardiac output. | Evaluations at 2 time points; when MAP is set to 65 and 95 mmHg. The evaluations are separated by approximately 30-60 min.
  Change in cardiac output [l/min] as evaluated by Swan Ganz catheter when MAP is set to 65 and 95 mmHg.
Change in cerebral oxygenation by near-infrared spectroscopy. | Evaluations at 2 time points; when MAP is set to 65 and 95 mmHg. The evaluations are separated by approximately 30-60 min.
  Change in cerebral oxygenation [%] as evaluated by near-infrared spectroscopy when MAP is set to 65 and 95 mmHg.
Change in pupillometry. | Evaluations at 2 time points; when MAP is set to 65 and 95 mmHg. The evaluations are separated by approximately 30-60 min.
  Change in pupil size and light reaction [mm and %] as evaluated by Neuroptics NPi-200 pupillometry when MAP is set to 65 and 95 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Niels D Olesen, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-07-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT05434910/SAP_000.pdf